CLINICAL TRIAL: NCT03996876
Title: Resolving Psychological Stress (RePS): a Mobile Health Application for Modifying Attention Bias to Threat in Post-traumatic Stress Disorder
Brief Title: Resolving Psychological Stress
Acronym: RePS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-10411
Record Dates: First submitted 2018-04-30; First posted 2019-06-25 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Post-Traumatic Stress Disorder; Alcohol Use Disorder
Keywords: Attention Bias Modification; PTSD; Digital Health; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a threat attention bias modification training or a neutral attention training.
Who Masked: Participant
Masking Description: Participants will be blind to the bias modification training they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Threat ABM Training (Active Comparator): Attention Bias Modification Training with threatening words
  Interventions: Device: RePS (Resolving Psychological Stress) - Threat ABM Training
- Neutral Attention Training (Placebo Comparator): Non-active version of ABM Training
  Interventions: Device: RePS (Resolving Psychological Stress) - Neutral Attention Training

INTERVENTIONS:
Device: RePS (Resolving Psychological Stress) - Threat ABM Training — This mobile "app" will aim to reduce neurobiological threat sensitivity with the ultimate goal of developing novel treatments for PTSD. The app can be used on an iPhone Operating System (iOS) compatible phone and involves a training program that aims to directly reduce threat sensitivity by modifying attention. The contents of the app will be the same for each user.
  Arms: Threat ABM Training
Device: RePS (Resolving Psychological Stress) - Neutral Attention Training — This app will be a placebo attention bias modification that will be used on an iOS compatible phone. The placebo will contain only neutral words.
  Arms: Neutral Attention Training

SUMMARY:
The investigators have developed a mobile app called Resolving Psychological Stress (REPS) to help alleviate symptoms of PTSD. The app will administer threat-related attention bias modification to individuals who have both a Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) diagnosis of PTSD (and meet at least one DSM-V criteria for threat sensitivity) and a DSM-V diagnosis of Alcohol Use Disorder. The aims of the study are to explore both the feasibility and acceptability of the app with it's users, and to explore the efficacy of the app at alleviating PTSD severity.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a highly disabling disorder that affects approximately 30 million people in the United States. New low-cost and accessible treatments for PTSD are desperately needed. Threat-related attention biases represent an important potential treatment target for PTSD. Such attention biases predict risk for PTSD following trauma exposure, and are thought to maintain symptoms of PTSD and other anxiety disorders. Research indicates that specific forms of computerized attention bias modification (ABM) are effective in reducing attention bias for threat as well as anxiety in patients with diverse anxiety disorders. The investigators have developed a mobile "app" called RePS (Resolving Psychological Stress) to administer threat-related ABM to patients with PTSD and Alcohol Use Disorder and have tested it in a laboratory-based pilot study of 19 people with PTSD. Preliminary data indicate that the app is highly acceptable to patients and that use of the app reduces attention bias for threat and PTSD symptom severity. The study aims are to examine the feasibility, acceptability and usability of app-based ABM; and determine the efficacy of app-based ABM in reducing attention bias and PTSD severity.

ELIGIBILITY:
Inclusion Criteria:

1. Must have current PTSD symptoms.
2. Must drink alcohol.

Exclusion Criteria:

1. Very recent or current trauma or trauma exposure.
2. Recent moderate or severe non-alcohol substance use disorder.
3. Active suicidality.
4. Lifetime history of schizophrenia or bipolar disorder I.
5. Medical conditions including seizure disorders, neurological disorders, moderate or severe head injury, systemic illness affecting nervous system function, heart defect, or medically unstable injuries.
6. Recent or planned change in psychotherapeutic treatment for PTSD or other psychiatric symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aoife S O'Donovan, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Aoife O'Donovan, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Threat ABM Training | Neutral Attention Training
Started | 14 | 14
Completed | 12 | 10
Not Completed | 2 | 4
Not completed — Incomplete Data | 2 | 4

BASELINE CHARACTERISTICS:
Population: Analyses of baseline characteristics have been conducted on the 28 participants that enrolled in the study.
Groups:
- Threat ABM Training; Neutral Attention Training: All participants used the same REPS app to complete their training. At the end of their training they answered general questions about the app that did not pertain to the specific type of training they received.
- Total: Total of all reporting groups
Arm/Group | Threat ABM Training | Neutral Attention Training | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.57 (9.25) | 39.30 (11.57) | 44 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 10 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Hawaiian or other Pacific Islander | 0 | 0 | 0
  Hispanic/Latinx | 0 | 2 | 2
  African American/Black | 2 | 5 | 7
  Caucasian/European American | 9 | 4 | 13
  Other | 0 | 0 | 0
  More than one ethnicity | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
PTSD Checklist-5 (PCL-5) Score [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 assesses the presence and severity of 20 different symptoms posttraumatic stress disorder (PTSD). Each of the 20 items is scored on a severity range of 0 (not at all) to 4 (extremely), for a final score range of 0-80. A score of 33 and above is indicative of clinically significant PTSD symptoms. Higher scores indicate worse PTSD symptom severity. Population: 1 participant did not complete the PCL at baseline.
  units on a scale
    number analyzed (Participants) | 14 | 13 | 27
    (all) | 36.07 (17.17) | 37.62 (20.99) | 36.81 (18.75)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms Using PTSD Checklist-5 (PCL-5) at Baseline and 15 Days
Description: The PTSD Checklist-5 (PCL- 5) was administered via the mobile application to assess changes in PTSD symptoms. The PCL-5 is a well validated and widely used structured 20-item diagnostic interview for assessing symptomology of PTSD corresponding to a DSM-5 diagnosis. PCL scores range from 0-80, with a score of 33 or above indicating clinically significant PTSD symptoms. Participants were asked about the severity of symptoms over the past week.
Time Frame: 15 days apart
Population: All participants used in analyses completed at least 16/20 items of the PCL-5 (total 20 items) on both Day 1 (Pre) and Day 15 (Post).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Threat ABM Training | Neutral Attention Training
Number analyzed (Participants) | 12 | 10
units on a scale
  Pre PCL Score | 33.2 (16.1) | 36.6 (20.9)
  Post PCL Score | 31.2 (15.8) | 28.2 (21.9)
Statistical Analysis 1: Comparison: Threat ABM Training vs Neutral Attention Training; Test type: Superiority — Given the relatively small sample size, results of our inferential statistical tests should be interpreted with caution; p = 0.322, ANOVA — The a priori threshold for statistical significance was set at 0.05; We conducted a two-way mixed ANOVA with intervention as the between-subjects and time as the within-subjects variable; F Statistic = 1.032 — The F Statistic reported is for the interaction between Intervention and Time

2. Primary Outcome: Differences in Heart Rate Variability (HRV) During a Threat Sensitivity Computerized Task
Description: Participants will perform computerized tasks designed to assess threat sensitivity. The task contains three different "threat" conditions, regarding the possibility of receiving a small, electric shock via an electrode on the hand (shock level is set by the participant). The three conditions are: shock not possible, shock possible, and shock may be possible. HRV is measured during all conditions and differences between the three conditions are scored.
Time Frame: 15 days apart
Population: Due to technical difficulties, we were unable to calculate heart rate variability for the participants in this study. Thus, HRV data was not collected in this study.
Arm/Group | Threat ABM Training | Neutral Attention Training
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rating of the Resolving Psychological Stress (Reps) Mobile Application on a Five-Point Scale for Multiple Feasibility and Acceptability Items After the Intervention, at 15 Days
Description: A usability assessment questionnaire was administered with multiple feasibility and acceptability questions regarding the REPS Mobile Application (Ease of use, Convenience, Enjoyment, Comfort with the app and Overall satisfaction). The responses were measured on a Five-Point Scale with 1 meaning "Not at all" and 5 meaning "Very much"." Analyses included all participants that completed the usability assessment questionnaire.
Time Frame: 15 days
Population: Analyses included all participants that completed the usability assessment questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Threat ABM Training | Neutral Attention Training
Number analyzed (Participants) | 12 | 10
score on a scale
  Ease of use | 4.56 (0.74) | 4.52 (0.90)
  Convenience | 4.02 (1.06) | 3.92 (1.16)
  Enjoyable | 3.29 (1.13) | 3.18 (1.22)
  Comfort with the app | 4.44 (0.80) | 4.41 (0.83)
  Overall satisfaction | 4.17 (0.87) | 4.05 (1.02)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the duration of participation which lasted eight weeks.
Arm/Group | Threat ABM Training | Neutral Attention Training
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

LIMITATIONS AND CAVEATS:
Sample size is limited and results should be interpreted cautiously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03996876/Prot_SAP_000.pdf